CLINICAL TRIAL: NCT06879015
Title: Tension Band Plate (TBP) vs Percutaneous Epiphysiodesis by Transphyseal Screw (PETS) in Coronal Angular Knee Deformities in Children: a Randomized Controlled Study
Brief Title: Plate vs. Screw for Guided Growth in Coronal Knee Deformities
Acronym: PETS vs TBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abdelghany Shazly, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-2025-201192
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Epiphysiodesis; Bone Malalignment; Lower Extremity Deformities, Congenital; Genu Varum; Genu Valgum
Keywords: Guided Growth; Growth Modulation; Tension Band Plate; Percutaneous Epiphysiodesis by Transphyseal Screw
MeSH Terms: conditions — Bone Malalignment; Lower Extremity Deformities, Congenital; Genu Varum; Genu Valgum | interventions — tributyl phosphate; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two groups, each receiving one of the two interventions (Tension Band Plate or Percutaneous Epiphysiodesis by Transphyseal Screw).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tension Band Plate (TBP) Group (Active Comparator): Participants in this group will undergo guided growth correction of coronal angular knee deformities using the Tension Band Plate (TBP) technique. A non-locking 8-plate is placed extraperiosteally across the growth plate with two screws to modulate bone growth gradually. This technique allows controlled correction without permanently damaging the physis and is commonly used for treating genu valgum and genu varum.
  Interventions: Procedure: Tension Band Plate (TBP) Surgery
- Percutaneous Epiphysiodesis by Transphyseal Screw (PETS) Group (Active Comparator): Participants in this group will undergo guided growth correction using Percutaneous Epiphysiodesis by Transphyseal Screw (PETS). This involves inserting a partially threaded cannulated screw across the growth plate to slow down growth on one side of the bone, achieving gradual angular correction. PETS is a minimally invasive alternative to TBP and has been associated with faster correction rates.
  Interventions: Procedure: Percutaneous Epiphysiodesis by Transphyseal Screw (PETS) Surgery

INTERVENTIONS:
Procedure: Tension Band Plate (TBP) Surgery — A guided growth procedure in which a non-locking 8-plate is placed extraperiosteally across the physis (growth plate) with two screws, one in the epiphysis and one in the metaphysis. This allows for gradual correction of coronal angular deformities without causing permanent growth arrest.
  Other Names: Guided Growth with Tension Band Plate; Extraperiosteal Growth Modulation with 8-Plate; Temporary Hemi-epiphysiodesis with Tension Band Plate; 8-Plate Hemi-epiphysiodesis
  Arms: Tension Band Plate (TBP) Group
Procedure: Percutaneous Epiphysiodesis by Transphyseal Screw (PETS) Surgery — A minimally invasive procedure in which a partially threaded cannulated screw is inserted across the growth plate (transphyseal) to slow growth on one side of the bone. This technique allows for gradual correction of genu valgum and genu varum.
  Other Names: Transphyseal Screw Epiphysiodesis; Growth Modulation with Transphyseal Screw; Minimally Invasive Epiphysiodesis with Screw
  Arms: Percutaneous Epiphysiodesis by Transphyseal Screw (PETS) Group

SUMMARY:
The goal of this clinical trial is to compare two surgical techniques, Tension Band Plate (TBP) and Percutaneous Epiphysiodesis by Transphyseal Screw (PETS), in children with coronal angular knee deformities.

The main questions it aims to answer are:

* Which technique provides better correction of coronal knee deformities?
* Are there differences in complication rates or recovery times between TBP and PETS?

Participants will:

* Undergo either TBP or PETS surgery for knee deformity correction.
* Attend follow-up visits for radiographic and clinical evaluations.

Researchers will compare TBP and PETS groups to see if one method leads to better deformity correction and fewer complications.

DETAILED DESCRIPTION:
Genu varum and genu valgum are common lower limb deformities observed in children and adolescents. These conditions often require guided growth techniques for correction. One widely accepted approach for modulating growth and gradually correcting these deformities is temporary Hemi-epiphysiodesis. The two most commonly used techniques for this purpose are the Tension Band Plate (TBP) e.g. Eight-Plate and Percutaneous Epiphysiodesis using Transphyseal Screws (PETS). While both methods have proven effective, there remains ongoing debate about their relative efficacy, safety, and long-term outcomes.

The TBP technique, introduced as a less invasive method of guided growth, involves placing a non-locking plate and screws across the growth plate on one side allowing controlled correction without permanent damage to the physis.

Studies have demonstrated its effectiveness in treating angular deformities with a lower risk of growth plate closure, but concerns remain regarding implant migration, breakage, and rebound deformity post-removal. Conversely, PETS offers a minimally invasive alternative where transphyseal screws modulate growth without requiring plate fixation. Some studies suggest PETS may provide more rapid correction with fewer complications, while others highlight the potential risk of premature physeal closure, which could lead to limb length discrepancies.

Despite the widespread use of both techniques, there is limited high-quality comparative data to determine the superior method in terms of correction rate, complication profile, and long-term functional outcomes. A randomized controlled study comparing TBP and PETS is essential to establish evidence-based guidelines, optimize patient outcomes, and refine surgical decision-making in the management of genu varum and genu valgum. Our novel introduction of the Bone-Length Adjusted Correction Rate as a new criterion will further enhance the measurement of effectiveness for these interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents beyond the age of physiological varus/valgus correction (i.e., typically ≥4 years for genu varum and ≥7 years for genu valgum) with Mechanical Axis Deviation (MAD) in lower limbs and abnormal joint orientation angles, in the coronal plane either femoral or tibial.
2. Open physis (growth plate) on radiographs and at least one year of growth remaining before age of skeletal maturity (typically ≤14 years in females, ≤16 years in males).

Exclusion Criteria:

1. Sick Physis as in Blount's disease stages III-V or any partial or total physeal arrest caused by trauma, inflammation or neoplasia.
2. Uncorrectable systemic disorders affecting bone growth and alignment, including but not limited to:

   i- Severe metabolic disorders (e.g., advanced rickets, hypophosphatasia, mucopolysaccharidoses) ii- Uncontrolled endocrine disorders (e.g., untreated hypothyroidism, growth hormone abnormalities) iii- Severe connective tissue disorders (e.g., osteogenesis imperfecta, advanced Ehlers-Danlos syndrome) iv- Chronic inflammatory or hematologic conditions that impair bone growth (e.g., severe juvenile idiopathic arthritis, advanced sickle cell disease)

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Bone-Length Adjusted Angular Correction Rate (BLAACR) | Measured at 3-month intervals until clinical correction is achieved, up to 12 months
  The Bone-Length Adjusted Angular Correction Rate (BLAACR) measures the effectiveness of guided growth correction by normalizing the angular correction rate based on limb growth. This method reduces bias in comparing the Tension Band Plate (TBP) and Percutaneous Epiphysiodesis by Transphyseal Screw (PETS) by accounting for variations in growth rate among participants. The formula is: BLAACR = (Change in Angular Deformity) / (Increase in Bone Length), where: -- Change in Angular Deformity = Initial Angle - Final Angle
  * Increase in Bone Length = Initial Bone Length - Final Bone Length

SECONDARY OUTCOMES:
Angular Correction Rate (Degrees/Month) | Measured at 3-month intervals until clinical correction is achieved, up to 12 months
  Measures the rate of angular deformity correction over time without adjusting for bone growth. This is calculated as: (Initial Angle - Final Angle) / Total Months of Follow-up.
Complications (Pain, Infection, Hardware Migration/Breakage) | Evaluated at each follow-up visit (3, 6, 9, 12 months)
  Assess the frequency and severity of complications related to TBP and PETS, including post-operative pain (measured using a visual analog scale), surgical site infections, implant migration, and hardware failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janarv PM, Wikstrom B, Hirsch G. The influence of transphyseal drilling and tendon grafting on bone growth: an experimental study in the rabbit. J Pediatr Orthop. 1998 Mar-Apr;18(2):149-54. PMID 9531394
- [Background] Tirta M, Hjorth MH, Jepsen JF, Kold S, Rahbek O. Staples, tension-band plates, and percutaneous epiphysiodesis screws used for leg-length discrepancy treatment: a systematic review and proportional meta-analysis. Acta Orthop. 2024 Jul 18;95:415-424. doi: 10.2340/17453674.2024.41104. PMID 39023429
- [Background] Schoenleber SJ, Iobst CA, Baitner A, Standard SC. The biomechanics of guided growth: does screw size, plate size, or screw configuration matter? J Pediatr Orthop B. 2014 Mar;23(2):122-5. doi: 10.1097/BPB.0000000000000026. PMID 24322536
- [Background] Ilharreborde B, Gaumetou E, Souchet P, Fitoussi F, Presedo A, Pennecot GF, Mazda K. Efficacy and late complications of percutaneous epiphysiodesis with transphyseal screws. J Bone Joint Surg Br. 2012 Feb;94(2):270-5. doi: 10.1302/0301-620X.94B2.27470. PMID 22323699
- [Background] Park BK, Kim HW, Park H, Lee SK, Park KB. Natural behaviours after guided growth for idiopathic genu valgum correction: comparison between percutaneous transphyseal screw and tension-band plate. BMC Musculoskelet Disord. 2022 Dec 3;23(1):1052. doi: 10.1186/s12891-022-05996-1. PMID 36461004
- [Background] Shapiro G, Adato T, Paz S, Shrabaty T, Ron L, Simanovsky N, Zaidman M, Goldman V. Hemiepiphysiodesis for coronal angular knee deformities: tension-band plate versus percutaneous transphyseal screw. Arch Orthop Trauma Surg. 2022 Jan;142(1):105-113. doi: 10.1007/s00402-020-03602-4. Epub 2020 Sep 21. PMID 32959086
- [Background] Eastwood DM, Sanghrajka AP. Guided growth: recent advances in a deep-rooted concept. J Bone Joint Surg Br. 2011 Jan;93(1):12-8. doi: 10.1302/0301-620X.93B1.25181. PMID 21196537
- [Background] Stevens PM, Klatt JB. Guided growth for pathological physes: radiographic improvement during realignment. J Pediatr Orthop. 2008 Sep;28(6):632-9. doi: 10.1097/BPO.0b013e3181841fda. PMID 18724199
- [Background] Khoury JG, Tavares JO, McConnell S, Zeiders G, Sanders JO. Results of screw epiphysiodesis for the treatment of limb length discrepancy and angular deformity. J Pediatr Orthop. 2007 Sep;27(6):623-8. doi: 10.1097/BPO.0b013e318093f4f4. PMID 17717460
- [Background] Boero S, Michelis MB, Riganti S. Use of the eight-Plate for angular correction of knee deformities due to idiopathic and pathologic physis: initiating treatment according to etiology. J Child Orthop. 2011 Jun;5(3):209-16. doi: 10.1007/s11832-011-0344-4. Epub 2011 May 12. PMID 22654982
- [Background] Metaizeau JP, Wong-Chung J, Bertrand H, Pasquier P. Percutaneous epiphysiodesis using transphyseal screws (PETS). J Pediatr Orthop. 1998 May-Jun;18(3):363-9. PMID 9600565